CLINICAL TRIAL: NCT00444613
Title: A Phase II/III Study in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E0302-J081-761
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2014-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis (ALS); motor neurons; muscular atrophy; Lou Gehrig's Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Muscular Atrophy | interventions — mecobalamin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- E0302 25 mg (Experimental)
  Interventions: Drug: E0302 (mecobalamin)
- E0302 50 mg (Experimental)
  Interventions: Drug: E0302 (mecobalamin)
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E0302 (mecobalamin) — Intramuscular injection, mecobalamin 25 mg twice a week for 3.5 years.
  Other Names: mecobalamin
  Arms: E0302 25 mg
Drug: E0302 (mecobalamin) — Intramuscular injection, mecobalamin 50 mg twice a week for 3.5 years.
  Other Names: mecobalamin
  Arms: E0302 50 mg
Drug: Placebo — Intramuscular injection, placebo twice a week for 3.5 years.
  Arms: 3

SUMMARY:
The purpose of this study is to investigate the efficacy and confirm the safety of E0302 in patients with Amyotrophic Lateral Sclerosis (ALS) by assessing changes in scores of survival rate and functional rating scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are able to submit written informed consent. If patients are duly capable of study consent but are unable to sign (or affix a seal) by themselves due to aggravation of disease condition, written informed consent can be obtained from a legally authorized representative who can sign on behalf of the patients after confirming the patients' agreement to study participation.
2. Patients who are aged 20 years or older at the time of obtaining informed consent.
3. Patients who have clinically definite ALS, clinically probable ALS, or clinically probable-laboratory supported ALS as specified in the revised El Escorial Airlie House diagnostic criteria.
4. Patients who are at stage 1 or 2 of the severity criteria for ALS.
5. Patients within 3-year elapsed time period from disease onset at the start of observation period.
6. Patients who can visit study site for out-patient treatment.

Exclusion Criteria:

1. Patients who underwent tracheostomy.
2. Patients who experienced non-invasive positive pressure ventilation.
3. Patients whose percent-predicted forced vital capacity (%FVC) is >=60%.
4. Patients with multiple disturbances of conduction detected by nerve conduction test.
5. Patients with neurological symptom(s) due to vitamin B12 deficiency.
6. Patients who initiated newly introduced riluzole therapy after starting the observation period. Or those who received dose escalation or resumed administration of riluzole therapy after previous down titration or discontinuation.
7. Patients with cognitive impairment.
8. Pregnant women or women with a possibility of becoming pregnant.
9. Patients or their partners who are not willing to use reliable contraception.
10. Patients with severe disease in the renal, cardiovascular, hematological, or hepatic system (severe disease will be judged referring to "Ministry of Health, Labor and Welfare" (MHLW) Drug Safety Dept. Notification No. 80, Drug Safety Classification Criteria for Severity of Adverse Drug Reaction by Medicinal Products, Grade 3).
11. Patients with malignant tumor.
12. Patients who participated in another clinical study within 12 weeks before starting the observation period.
13. Patients with present illness or history of drug allergy or severe allergic disease (anaphylactic shock).
14. Patients who are judged to be ineligible for study entry by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2007-04; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Survival rate | Every 3 months.
Functional rating scale. | Every 3 months.

SECONDARY OUTCOMES:
Manual Muscle Test (MMT) | Every 3 months.
Percent-predicted forced vital capacity (%FVC) | Every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kazunori Saeki, Study Director — Neuroscience Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (44):
- Japan (44):
  - Nagoya, Aichi-ken
  - Akita, Akita
  - Aomori, Aomori
  - Chiba, Chiba
  - Touon-shi, Ehime
  - Fukuoka, Fukuoka
  - Kitakyusyu-shi, Fukuoka
  - Fukushima, Fukushima
  - Maebashi, Gunma
  - Higashihiroshima-shi, Hiroshima
  - Miyoshi-shi, Hiroshima
  - Otake-shi, Hiroshima
  - Sapporo, Hokkaido
  - Kanazawa, Ishikawa-ken
  - Ichinoseki-shi, Iwate
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Nangoku-shi, Kochi
  - Kyoto, Kyoto
  - Tsu, Mie-ken
  - Sendai, Miyagi
  - Watari-gun, Miyagi
  - Nagano, Nagano
  - Higashisonogi-gun, Nagasaki
  - Kashiwazaki-shi, Niigata
  - Niigata, Niigata
  - Tsukubo-gun, Okayama-ken
  - Ginowan-shi, Okinawa
  - Toyonaka-shi, Osaka
  - Hasuda-shi, Saitama
  - Saitama-shi, Saitama
  - Ōtsu, Shiga
  - Hamamatsu, Shizuoka
  - Shizuoka, Shizuoka
  - Shimotsuke-shi, Tochigi
  - Tokushima, Tokushima
  - Yoshinogawa-shi, Tokushima
  - Bunkyo-ku, Tokyo
  - Kodaira-shi, Tokyo
  - Ōta-ku, Tokyo
  - Wakayama, Wakayama
  - Yonezawa-shi, Yamagata
  - Shimonoseki-shi, Yamaguchi
  - Yanai-shi, Yamaguchi

REFERENCES:
- [Derived] Kaji R, Imai T, Iwasaki Y, Okamoto K, Nakagawa M, Ohashi Y, Takase T, Hanada T, Shimizu H, Tashiro K, Kuzuhara S. Ultra-high-dose methylcobalamin in amyotrophic lateral sclerosis: a long-term phase II/III randomised controlled study. J Neurol Neurosurg Psychiatry. 2019 Apr;90(4):451-457. doi: 10.1136/jnnp-2018-319294. Epub 2019 Jan 13. PMID 30636701
- [Derived] Ikeda K, Iwasaki Y, Kaji R. Neuroprotective effect of ultra-high dose methylcobalamin in wobbler mouse model of amyotrophic lateral sclerosis. J Neurol Sci. 2015 Jul 15;354(1-2):70-4. doi: 10.1016/j.jns.2015.04.052. Epub 2015 May 8. PMID 25982504